CLINICAL TRIAL: NCT06168162
Title: Effect of Individualized High Positive End-expiratory Pressure on Postoperative Pulmonary Rate in Laparoscopic Bariatric Surgeries
Brief Title: Effect of Individualized PEEP on Postoperative Pulmonary Complication in Bariatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD259/2023
Record Dates: First submitted 2023-11-04; First posted 2023-12-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Mechanical Ventilation Pressure High; Bariatric Surgery Candidate
Keywords: ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- titrate PEEP (Experimental): individulaized PEEP starting 7cmH2O titrated to best static compliance (Cstat) ranging from 50 -100 cmH2O
  Interventions: Other: titated PEEP to best static compliance
- standard (Active Comparator): standard PEEP of 5 cmH2O
  Interventions: Other: titated PEEP to best static compliance

INTERVENTIONS:
Other: titated PEEP to best static compliance — the Intraoperative PEEP will be titrated to best static compliance for each patient

SUMMARY:
Ventilation with low tidal volume and high PEEP (positive end expiratory pressure) has been shown to improve oxygenation in patients with ARDS (acute respiratory distress syndrome). In obese patients undergoing laparoscopic bariatric surgeries, the risk of postoperative pulmonary complications (PPCs) increases significantly with general anesthesia. Previous studies have shown that protective lung ventilation strategies could improve intraoperative oxygenation and lung mechanics.

In this study would compare the effect of optimum individualized high PEEP versus standard PEEP - on postoperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for participation if the met the following criteria

  * Age between 18 and 60 years old.
  * Body mass index > 40
  * Laparoscopic bariatric elective surgery under general anesthesia.
  * ARISCAT (Assess Respiratory Risk in Surgical Patients in Catalonia) score ≥ 45 . ARISCAT score is a clinically practical seven-factor scoring system to assess the risk of a composite PPC.

Exclusion Criteria:

* Previous lung surgery
* ASA status III or IV.
* Moderate to severe obstructive or restrictive lung disease .
* Persistant intraoperative hemodynamic instability .
* Need for postoperative mechanical ventilation

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complication | postoperative 10 days after surgery
  pneumonia-atelactasis-bronchospasm-respiratory failure

SECONDARY OUTCOMES:
Pulmonary functions test | postoperative 1st , 3rd and 5th day
  This test includes these values :FVC (forced vital capacity ) FEV1( forced expiratory volume in one sec ) FEV1% and FVC%

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the results